CLINICAL TRIAL: NCT01554943
Title: Late Cardiac Evaluation of the Three Arm Belgian Trial A Phase III Randomized Trial Involving Node-positive Early Breast Cancer Patients With a Long Median Follow-up (~ 15 Years)
Brief Title: Late Cardiac Evaluation of the Three Arm Belgian Trial Involving Node-positive Early Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Collaborators: Centre Hospitalier Universitaire de Tivoli (Other); Clinique Sainte Elisabeth (Unknown); Centre Hospitalier Jolimont-Lobbes (Unknown); Réseau Hospitalier Médecine Sociale d'Ath (Unknown); Hôpital de Braine-l'Alleud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CE1740
Record Dates: First submitted 2012-03-08; First posted 2012-03-15 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Breast Cancer
Keywords: CMF; HEC; EC; node positive; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CMF (Active Comparator): adjuvant standard CMF given from 1988 to 1996
  Interventions: Other: cardiac MRI
- EC (Experimental): Adjuvant EC chemotherapy given from 1988 to 1996
  Interventions: Other: cardiac MRI
- HEC (Experimental): High dose epirubicin (HEC) given from 1988 to 1996
  Interventions: Other: cardiac MRI

INTERVENTIONS:
Other: cardiac MRI — Patients will be submitted to extensive cardiac evaluation several years after completion of adjuvant chemotherapy

SUMMARY:
Late Cardiac Evaluation of the Three Arm Belgian Trial A phase III randomized trial involving node-positive early breast cancer patients with a long median follow-up (~ 15 years)

OBJECTIFS

Primary:

• To compare the incidence of late cardiac events between anthracycline and non-anthracycline chemotherapy given to node-positive breast cancer patients in the Belgian three arm randomized clinical trial

Secondary:

* To compare the late incidence of cardiac events between higher and lower dose anthracycline treated node-positive breast cancer patients;
* To compare anthracyclines (higher and lower doses) and non-anthracycline chemotherapy for:
* left ventricular diastolic function assessed by Echo
* exercise capacity assessed by 6-minute walk test (6MWT)
* cardiac morphology (myocardial inflammation or injury, fibrosis, LVEF) assessed by MRI
* serum cardiac biomarkers (BNP and TNT)
* patient-reported cardiac symptoms
* patient-reported cardiac symptoms assessed by QOL questionnaires are associated with subclinical findings on LVEF assessment
* cognitive function, functional autonomy, and psychological distress

DETAILED DESCRIPTION:
The primary objective of this study is to compare the incidence of cardiac events [(defined as asymptomatic systolic dysfunction (LVEF < 50%, asymptomatic NYHA I) or symptomatic heart failure NYHA class II-IV either by Echo and/or by clinical exam (LVEF < 50% and heart failure symptoms)] between anthracycline and non-anthracycline chemotherapy treated node-positive breast cancer patients in a long-term follow-up. We will define a binary status for each patient: no cardiac event / one or more cardiac events. Analysis of the primary endpoint will involve a comparison of the CMF-treated patients versus the pooled anthracycline treated patients (EC and HEC). If a significant difference is detected, all paired comparisons will also be performed for the primary endpoint (CMF versus EC, CMF versus HEC, EC versus HEC).

ELIGIBILITY:
Inclusion Criteria:

* Alive, free of any recurrence, Not lost to follow-up
* Last workup should be no older than 1 year to exclude relapses. If this is older than 1 year, a new workup (PE, blood tests and MMG) will be performed prior to the entry in this study
* Patients previously diagnosed with CHF who are free of recurrence will also be invited to participate, if there is no contra-indication
* Patients should be able to perform the prescribed assessments

Exclusion Criteria:

* Death
* Breast cancer recurrence
* Unwilling to perform exams as per protocol

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2010-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Late cardiac toxicity | Exams will be performed only once, which will take place several years after the completion of chemotherapy (up to 15 years)
  The primary objective of this study is to compare the incidence of cardiac events [(defined as asymptomatic systolic dysfunction (LVEF < 50%, asymptomatic NYHA I) or symptomatic heart failure NYHA class II-IV either by Echo and/or by clinical exam (LVEF < 50% and heart failure symptoms)] between anthracycline and non-anthracycline chemotherapy. Analysis of the primary endpoint will involve a comparison of the CMF-treated patients versus the pooled anthracycline treated patients (EC and HEC).

SECONDARY OUTCOMES:
Late cardiac and cognitive toxicity | Exams will be performed only once, which will take place several years after the completion of chemotherapy (up to 15 years)
  * To compare the late incidence of cardiac events between higher and lower dose anthracycline treated node-positive breast cancer patients;
  * To compare anthracyclines (higher and lower doses) and non-anthracycline chemotherapy for: LVEF assessed by Echo; exercise capacity assessed by 6-minute walk test; cardiac morphology assessed by MRI; serum cardiac biomarkers; patient-reported cardiac symptoms assessed by QOL questionnaires; cognitive function, functional autonomy, and psychological distress

CONTACTS AND LOCATIONS:
Overall Officials: Evandro de Azambuja, MD, PhD, Principal Investigator — Jules Bordet Institute
Locations (1):
- Jules Bordet Institute, Brussels, Belgium

REFERENCES:
- [Background] Piccart MJ, Di Leo A, Beauduin M, Vindevoghel A, Michel J, Focan C, Tagnon A, Ries F, Gobert P, Finet C, Closon-Dejardin MT, Dufrane JP, Kerger J, Liebens F, Beauvois S, Bartholomeus S, Dolci S, Lobelle JP, Paesmans M, Nogaret JM. Phase III trial comparing two dose levels of epirubicin combined with cyclophosphamide with cyclophosphamide, methotrexate, and fluorouracil in node-positive breast cancer. J Clin Oncol. 2001 Jun 15;19(12):3103-10. doi: 10.1200/JCO.2001.19.12.3103. PMID 11408507
- [Background] de Azambuja E, Paesmans M, Beauduin M, Vindevoghel A, Cornez N, Finet C, Ries F, Closon-Dejardin MT, Kerger J, Gobert P, Focan C, Tagnon A, Dolci S, Nogaret JM, di Leo A, Piccart-Gebhart MJ. Long-term benefit of high-dose epirubicin in adjuvant chemotherapy for node-positive breast cancer: 15-year efficacy results of the Belgian multicentre study. J Clin Oncol. 2009 Feb 10;27(5):720-5. doi: 10.1200/JCO.2008.17.2155. Epub 2008 Dec 22. PMID 19103732
- [Derived] de Azambuja E, Ameye L, Diaz M, Vandenbossche S, Aftimos P, Bejarano Hernandez S, Shih-Li C, Delhaye F, Focan C, Cornez N, Vindevoghel A, Beauduin M, Lemort M, Paesmans M, Suter T, Piccart-Gebhart M. Cardiac assessment of early breast cancer patients 18 years after treatment with cyclophosphamide-, methotrexate-, fluorouracil- or epirubicin-based chemotherapy. Eur J Cancer. 2015 Nov;51(17):2517-24. doi: 10.1016/j.ejca.2015.08.011. Epub 2015 Aug 27. PMID 26321502